CLINICAL TRIAL: NCT04759612
Title: Is Self-action Observation More Effective Than Observing Another Person's Action During Upper Extremity Functions?
Brief Title: Is Self-action Observation More Effective Than Observing Another Person's Action?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Yusuf EMUK, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Katip Celebi University
Record Dates: First submitted 2021-02-05; First posted 2021-02-18 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Action Observation (s-AO Group) (Experimental): Participants will watch their own actions during an upper extremity functionality test.
  Interventions: Other: Action Observation
- Action Observation (AO Group) (Experimental): Participants will watch another person's actions during an upper extremity functionality test.
  Interventions: Other: Action Observation

INTERVENTIONS:
Other: Action Observation — Participants will watch an upper extremity functionality test.

SUMMARY:
The aim of the study is to compare the possible effects of self-action observation and observation of another person's action on upper extremity functionality, cognitive functions and reaction times.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* willingness

Exclusion Criteria:

* any kind of neurological or musculoskeletal problems
* sight problems
* pain in the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in upper extremity functionality | The outcome will be assessed at baseline and immediately after the intervention.
  Jebsen-Taylor Hand Function Test will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No